CLINICAL TRIAL: NCT00944944
Title: A Pilot Study Using the Gynecologic Cancer Lymphedema Questionnaire as a Clinical Care Tool to Identify Lower Extremity Lymphedema
Brief Title: Gynecologic Cancer Lymphedema Questionnaire as a Clinical Care Tool to Identify Lower Extremity Lymphedema
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Richard Barakat, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 09-077
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2010-02-01 (Estimated); Status verified 2010-01

CONDITIONS: Ovarian Cancer; Uterine Cancer; Vaginal Cancer; Lymphedema
Keywords: CORPUS UTERI,; ENDOMETRIUM; FALLOPIAN TUBE; OVARY; VAGINA; Lymphedema; Questionnaire; Quality of Life; 09-077; Fallopian Tubes
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Neoplasms; Vaginal Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Gyn Pts with lymphedema
  Interventions: Behavioral: GCLQ lymphedema symptom assessment questionnaire
- Gyn Pts without Lymphedema
  Interventions: Behavioral: limb volume measurements and GCLQ lymphedema symptom assessment questionnaire

INTERVENTIONS:
Behavioral: limb volume measurements and GCLQ lymphedema symptom assessment questionnaire — Upon obtaining consent, the participants without a history of lower extremity lymphedema will be asked to undergo limb volume measurements to ensure the accuracy of group assignment to the nonlymphedema group. Participants will then be asked to complete the one time GCLQ lymphedema symptom assessment questionnaire. The survey tool and Limb volume (LV) data and feedback from participants about the GCLQ will be collected. We expect the study survey to take approximately 5-10 minutes to complete and 5-10 minutes to collect LV data.
  Other Names: After completion of the GCLQ lower extremity lymphedema assessment tool, participants will be asked; to provide feedback about their satisfaction with and the feasibility of using this brief assessment tool!; screening mechanism to identify lymphedema symptoms in the clinical care setting.
  Groups: Gyn Pts without Lymphedema
Behavioral: GCLQ lymphedema symptom assessment questionnaire — The gynecologic cancer survivors with lymphedema group will have documented lower extremity lymphedema. Participants will be asked to complete a one time assessment, the Gynecologic Cancer Lymphedema Questionnaire to identify lower extremity lymphedema symptoms in gynecologic cancer survivors. They will also be asked to provide feedback about their satisfaction with and the feasibility of the GCLQ as a brief assessment tool that could be used in the clinical care setting.
  Groups: Gyn Pts with lymphedema

SUMMARY:
The purpose of this study is to evaluate if the Gynecologic Cancer Lymphedema Questionnaire (GCLQ) truly detects symptoms or signs of lower extremity lymphedema in patients with diagnosed lower extremity lymphedema. Lymphedema is a chronic condition in which fluid accumulates in the tissues of the body. Many cancer survivors are living with discomfort and changes in their activities due to limb swelling following cancer treatment. If the GCLQ is able to do detect signs and symptoms of lymphedema, the investigators hope to use it as a tool in the clinical care setting to help identify women at risk for or with lymphedema. In the future, this could improve clinical care through the use of a more simple and feasible way to identify lower extremity lymphedema than measuring limbs.

ELIGIBILITY:
Inclusion Criteria:

* Study group of Gynecologic cancer survivors with Lymphedema
* Documented lower extremity lymphedema
* History of a primary diagnosis of gynecologic cancer (vulvar, cervical and uterine only)
* History of surgery for gynecologic cancer including lymph node removal
* No evidence of disease or active treatment
* At least 21 years of age
* Able and willing to provide informed consent
* English fluency Comparison Group of Gynecologic Cancer Survivors without Lymphedema
* No history of lower extremity lymphedema or presence of lymphedema confirmed by limb volume measurements at the time of study participation
* History of a primary diagnosis of gynecologic cancer (vulvar, cervical and uterine only)
* History of surgery for gynecologic cancer including lymph node removal
* No evidence of disease or active treatment
* At least 21 years of age
* Able and willing to provide informed consent
* English fluency

Exclusion Criteria:

* Inability to participate in an informed consent process
* Patients with a psychiatric disorder precluding response to the survey

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential GYN research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine if the Gynecologic Cancer Lymphedema Questionnaire (GCLQ)tools detects lower extremity lymphedema symptoms in gynecologic cancer survivors & if it is a feasible assessment tool which can be used in the clinical care setting. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Barakat, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm